CLINICAL TRIAL: NCT04861766
Title: A Controlled, Prospective, Randomized, Multi-Center, Subject and Evaluator-Blinded Study of the Safety and Effectiveness of STYLAGE® L Versus Restylane® for Correction of Moderate and Severe Nasolabial Folds in Chinese Adults
Brief Title: Safety and Effectiveness of STYLAGE® L for Correction of Moderate and Severe Nasolabial Folds in Chinese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIV-STYL-L-01
Record Dates: First submitted 2021-04-26; First posted 2021-04-27 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Aging; Skin Wrinkling
Keywords: hyaluronic acid; Nasolabial Folds; Dermal filler

STUDY DESIGN:
Intervention Model Description: A Controlled, Prospective, Randomized, Multi-Center, Subject and Evaluator-Blinded Study
Who Masked: Participant, Outcomes Assessor
Masking Description: The identity of individual investigation materials will remain unknown to the independent Blinded Evaluator and all subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group Stylage L ® (Experimental): Each subject will receive STYLAGE® L in both NLFs.
  STYLAGE® L will be injected in the NLFs by the Treating Investigator with optional touch-up injections on Month 1.
  Interventions: Device: STYLAGE® L
- Control group Active Comparator (Active Comparator): Each subject will receive the Active Comparator in both NLFs.
  Active Comparator will be injected in the NLFs by the Treating Investigator with optional touch-up injections on Month 1.
  Interventions: Device: Active Comparator

INTERVENTIONS:
Device: STYLAGE® L — Injection in both NLFs
  Arms: Treatment group Stylage L ®
Device: Active Comparator — Injection in both NLFs
  Arms: Control group Active Comparator

SUMMARY:
This is a safety and efficacy study of STYLAGE® Lin Chinese adults with Nasolabial Folds.

DETAILED DESCRIPTION:
This is a prospective, multi-center, parallel-group, subject and evaluator-blinded, randomized controlled trial to demonstrate the non-inferiority of the study device, STYLAGE® L, when compared to an active comparator for the correction of moderate and severe NLFs.

Subjects will randomly receive STYLAGE® L or the active comparator (ratio 1:1) injection in the NLFs at first visit on Day 0.

Proportion of subjects having a NLFs severity improvement (blinded evaluation), 6 months after treatment initiation will be assessed and compared between the two groups. This will also be done during the other visits (1, 3, 9 and 12 months after treatment initiation). Global aesthetic improvement according to blinded independent evaluator and subject, subjects' satisfaction, and safety parameters will also be assessed during the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged ≥ 18 years.
2. Chinese ethnicity.
3. Subjects who wanting to correct his/her nasolabial folds
4. Subjects with moderate to severe nasolabial folds (attaining grade 3 on both side or 4 on both side) in the WSRS of nasolabial fold, per assessment of the Blinded Evaluator.
5. Subjects willing to abstain from other facial plastic surgical or cosmetic procedures during the study period.
6. Subjects with realistic expectations who can understand and comply with the instructions and all visit schedule.
7. Women of childbearing potential (WOCBP) who agree contraception during the study period.
8. Subjects who voluntarily decided the participation of the study and signed the informed consent.
9. Being able to stand mild pain.

Exclusion Criteria:

1. Subjects who are contraindicated to augmentation with HA fillers
2. Subjects who had a history of keloid formation or hypertrophic scar
3. Subjects presenting a scar or skin disorder (i.e. active dermal disease [facial psoriasis, eczema, rosacea, perioral dermatitis, acne, herpes, etc], inflammation or an unhealed wound) below the level of the lower orbital rim that may confound the study evaluation
4. Has ever received semi-permanent fillers or permanent facial implants (eg, calcium hydroxyapatite, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafluoroethylene) anywhere below the inferior orbital rim, or is planning to be implanted with any of these products at any time during the study
5. Has undergone temporary dermal filler treatment (e.g., hyaluronic acid or collagen) below the inferior orbital rim within 12 months before enrollment or is planning to undergo such treatment during the study
6. Has undergone facial tissue augmentation with fat injections, botulinum toxin injections, mesotherapy, or cosmetic facial procedures (eg, facial liposuction, aesthetic surgery, face-lift, photomodulation, intense pulsed light, radio frequency, dermabrasion, laser or chemical peel, or other ablative procedures) below the inferior orbital rim within 6 months before enrollment or is planning to undergo any such treatment during the study
7. Subjects who has any history of severe multiple allergies or an allergy resulting in anaphylaxis, or an allergy to hyaluronic acid and/or one of the ingredients of the study products
8. Subject is pregnant or planning to be pregnant during the study period or lactating. Women of childbearing potential who have a positive pregnancy test result during screening. Women of childbearing potential who are unwilling to use effective birth control measures during the full course of the study
9. Subject suffering from a serious or progressive disease, which, in the Investigator's judgment, put the subject at undue risk for participation in this clinical trial (i.e. cancer or pre-cancer, immunocompromised, uncontrolled diabetes, epilepsy, severe cardio-cerebrovascular disease(s) (i.e. stroke, idiopathic aortic stenosis, aneurysm, hypertrophic obstructive cardiomyopathy, ischaemic heart disease, tachyarrhythmias, severe heart failure [classified as NYHA III-IV], etc), , etc.)
10. Subject having a history of cancer within 5 years
11. Subjects who received oral surgery (eg. tooth extraction, orthodontia or implantation) within 6 weeks before enrollment or is planning to undergo any of these procedures during the study
12. Subject has history or active autoimmune disease (e.g. inflammatory bowel disease), active or history of connective tissue disease (rheumatoid arthritis, scleroderma, and systemic lupus erythematosus)
13. Subjects with current or a history of hemorrhagic diseases
14. Subject who received chemotherapy, immunosuppressive agents, immunomodulatory therapy (e.g. monoclonal antibodies), systemic corticosteroids within 3 months (inhaled corticoids are allowed).
15. Subjects unlikely to achieve a meaningful aesthetic result with the prescribed dosage regimen of the study product per Investigator's judgement
16. Subjects who participated in other clinical trial within 30 days or who is in an exclusion period of one.
17. Subjects with uncontrolled hypertension (systolic blood pressure above 160mmHg or diastolic blood pressure above 100 mmHg at resting status), and/or significant liver (serum ALT or AST ≥2X the upper limit of the reference range), kidney (BUN, Urea or Cr≥1.5X the upper limit of the reference range), and/or blood coagulation (PT, or APTT, or INR> 20% of the reference range) disorders per judgement of the Investigator.
18. Current or a history of alcoholism, drug abuse, or drug dependence.
19. Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship
20. Subject with a past history of streptococcal disease (manifested by recurrent sore throat or acute rheumatic fever) or with an active infection to streptococcus
21. Has facial hair (e.g., beards, sideburns, etc.), piercing or tattoo in the area to be treated that would interfere with investigation assessments and create inconsistency in required investigation photography during the study period
22. Personnel of the study department, close relatives of the study department personnel (i.e. parents, children, siblings, or spouse), employees, or close relatives of employees at the Sponsor or CRO company.
23. Other conditions the Investigator considers inappropriate for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
WSRS improvement | Month 6
  Percentage of responders, defined by at least 1-point improvement from baseline 5-point WSRS, as measured by the Blinded Evaluator at 6 months after last treatment for both groups.

SECONDARY OUTCOMES:
WSRS improvement | 1, 3, 9, and 12 months
  Percentage of responders, defined by at least 1-point improvement from baseline 5-point WSRS, as measured by the Blinded Evaluator
GAIS assessment | 1, 3, 9, and 12 months
  Percentage of responders, defined by having "Improved", "Much improved" or "Very much improved" according to the Global Aesthetic Improvement Scale (GAIS), as assessed by the subject and the Treating Investigator
Subject satisfaction assessment | 1, 3, 6, 9, and 12 month
  Percentage of satisfied subjects on each question of the subject satisfaction assessment
Device performance | initial and touch up
  Results of device performance evaluation after the initial and touch-up injection, respectively, by the Treating Investigator for both groups.
Report of Adverse Event | Day 0, Month 1, Month 3, Month 6, Month 9, Month 12
  Product safety will be assessed by collection of local tolerability after each injection session, and Adverse Events (AEs) throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wu, Principal Investigator — Peking University First Hospital
Locations (8):
- China (8):
  - Beijing Hospital, Beijing, Dong Cheng District
  - SUN YAT-SEN Memorial Hospital, SUN YAT-SEN University, Guangzhou, Guangdong
  - Guangdong Second Provincial General Hospital, Guangzhou, Guangdong
  - Air Force Medical Center, PLA, Beijing, Haidian District
  - Peking University Third Hospital, Beijing, Haidian District
  - West China Hospital of Stomatology Sichuan University, Chengdu, Sichuan
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Peking University First Hospital, Beijing, Xicheng District